CLINICAL TRIAL: NCT01752192
Title: Tele-rehabilitation of Heart Patients
Brief Title: Teledi@Log - Tele-rehabilitation of Heart Patients
Acronym: Teledi@log
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: KMD (Unknown); International Business Machines (IBM) (Industry); Tunstall Healthcare (Unknown); Oscar Film (Unknown); Roche Pharma AG (Industry); SOS International (Unknown); Danish Heart Foundation (Other); Hjoerring Municipaility (Unknown); Frederikshavn Municipality (Unknown); Regionshospital Nordjylland (Other Government); Aalborg University Hospital (Other); University of Aarhus (Other); GP in the Municipalities of Hjoerring and Frederikshavn (Unknown); EIR (Empowering Industry and Research) (Other)
Responsible Party: Principal Investigator, Birthe Dinesen, Associate professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-20120051; N-20120051 (Other Grant/Funding Number: EIR Businesspark and cofinancing from partners)
Record Dates: First submitted 2012-12-12; First posted 2012-12-19 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure; Myocardial Infarction; Angina Pectoris; Coronary Stenosis; Mitral Valve Stenosis
Keywords: Rehabilitation; Telemedicine; Heart patients; Social media; Organisational aspects
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Angina Pectoris; Coronary Stenosis; Mitral Valve Stenosis | interventions — Blood Pressure Monitors

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telerehabilitation programme (Experimental): Telerehabilitation programme: Each patient will use a telehealth monitor and measure blood pressure, pulse and weight once or twice a week over a 3 months periods with the use of a blood pressure monitor and a weightscale connected to the monitor. The patients will also measure their steps daily by the use of a digital step-counter. The patients will be able to see their data in a personal health record on a tablet where they can share informations with healthcare professionals. The patient are also offered access to a portal called www.aktivehjerte.dk where they can find informations on rehabilitations topics in text, video and sound. The patients are randomised in block of different sizes to follow rehabilitation from hospital, healthcare center or a callcenter.
  Interventions: Device: Telerehabilitation programme
- Control group traditional rehabilitation (No Intervention): The control group of heart patients follow traditional rehabilitation activities for a period of 3 months.The patients are randomised in block of different sizes to follow rehabilitation from hospital, healthcare center or a callcenter.

INTERVENTIONS:
Device: Telerehabilitation programme — Telerehabilitation programme: Each patient in the intervention group will use a telehealth monitor. The patient will measure blood pressure, pulse and weight once or twice a week over a 3 months periode with the use of a blood pressure monitor and a weightscale connected to the monitor. The patients will also measure their steps daily by the use of a digital stepcounter. The patients will be able to see their data in a personal health record on a tablet where they can share informations with their GP, nurse and doctor at the hospital or healthcare center. The patient are also offered access to a portal called www.aktivehjerte.dk where they can find informations on rehabilitations topics in text, video and sound.
  Other Names: MyMedic (RTX 3370/71); Blood Pressure Monitor; Weight Scale; FitBit Zip(Stepcounter); Tablet(Samsung Galaxy Tab 2 10.1)
  Arms: Telerehabilitation programme

SUMMARY:
The idea behind the Teledi@log consortium is to develop tele-rehabilitation concepts and technologies so that all types of heart disease patients, regardless of degree of severity, can be offered individual, customized and coordinated tele-rehabilitation across sectors. The project is innovative, breaking new ground in relation to existing national and international research projects in the area. The Teledi@log consortium sees its major task as developing and testing scenarios which can lead to a more coherent rehabilitation for heart patients in areas such as patient training, organization across the boundaries of the health system and using tele-rehabilitation technology. The Teledi@log consortium seeks to develop new tele-rehabilitation concepts which bring the patient closer to the health system and thereby promote the heart patient's rehabilitation, giving the patient and their families a more active role via new tele-rehabilitation technologies.The hypothesis of the study is that heart patients participating in a telerehabilitation program will have a higher quality of life compared to heart patients following traditional rehabilitation activities.

DETAILED DESCRIPTION:
The aims of the research project are:

To assess the heart patients' and family members' needs for rehabilitation in the health system

To assess the need for coordination of the rehabilitation effort in the health system

To develop tele-rehabilitation concepts and technologies for heart patients, family members and health professionals in the health sector

To promote an early, rapid and effective rehabilitation of heart patients to improve their daily life and working life.

To prevent re-hospitalization of heart patients through a more individualized and differentiated rehabilitation effort using tele-rehabilitation technologies.

To conduct a randomized study of a tele-rehabilitation concept using tele-rehabilitation technologies and to assess the clinical, technical, organizational and health-economic effects.

ELIGIBILITY:
Inclusion Criteria:

* Women and men above 18 years
* Must have signed the "Informed Consent" document
* Must be able to understand study information
* Must live in Hjørring or Frederikshavn Kommune
* Must have mobile network
* Must be able to use IT or have a near person who can use IT
* Patients with clinical diagnosis of Heart Failure, Myocardial Infarction, Angina Pectoris, patients who have had Coronary-Artery Bypass Surgery.

Exclusion Criteria:

* Patients who, according to investigator, will not be able to participate in the study
* Lack of ability to speak and understand Danish
* Pregnancy or nursing
* Neurologic disease
* Use of wheelchair/lack of ability to walk
* Participation in other studies which can influence the outcomes of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Quality of life | At inclusion (baseline), change from baseline at 3, 6 and 12 months
  Quality of life is measured via the questionaire SF 36 (short form health survey) at baseline (at inclusion) and changes from baseline at 3, 6 and 12 months.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | At inclusion (baseline), change from baseline at 3, 6 and 12 months
  To measure the patients degree of anxiety and depression at baseline (inclusion), changes from baseline at 3, 6 and 12 months.
Self-determination | At inclusion (baseline), change from baseline at 3, 6 and 12 months
  Questionaires on self-determination will be used in order to get an impression of the patients perception on handling their disease at baseline(inclusion)and changes from baseline at 3, 6 and 12 months.
Health outcome EQ 5 | At inclusion (baseline), change from baseline at 3, 6 and 12 months
  To measure health outcome at baseline (inclusion, and changes from baseline at 3, 6 and 12 months.
Health economical evaluation | At inclusion (baseline), change from baseline at 3, 6 and 12 months
  An assessment of the economical perspective of the telerehabilitation programme will be performed at baseline (inclusion of patients) and changes from baseline at 3, 6 and 12 months.
Interorganizational aspects of a telerehabilitation programme | Cnanges during 2012-2014
  Interorganiszational aspect of the crosssectional telerehabilitation programme will be explored through observations and qualitative interviews with healthcare professionals at baseline (start of the study) and changes from baseline will be identified in October 2013.
Social media for telerehabilitation | Changes within 3 months
  Patients use of social media during an rehabilitation process will be explored through interviews at baseline (inclusion) and changes from baseline at 3, 6 and 12 months will be identified.

OTHER OUTCOMES:
Perception of health | At inclusion (baseline), changes from baseline at 3, 6 and 12 months
  To identify the patients feeling of their health during telerehabilitation
Steps taken | At inclusion (baseline) and changes from baseline will be indtified
  To measure steps taken with a step counter at baseline(inclusion) and Changes during 12 months
Qualitative perceptions of telerehabilitation | Changes within 3 months
  To explore patients perceptions of participating in a telerehabilitation program at baseline (incluion) and changes from baseline at 3, 6 and 12 months will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Birthe Dinesen, PhD, Principal Investigator — Aalborg University
Locations (2):
- Denmark (2):
  - Thoracic Ward, Aalborg University Hospital, Aalborg
  - Cardiology Ward Vendyssel Hospital, Hjørring

REFERENCES:
- [Result] Dithmer M, Rasmussen JO, Gronvall E, Spindler H, Hansen J, Nielsen G, Sorensen SB, Dinesen B. "The Heart Game": Using Gamification as Part of a Telerehabilitation Program for Heart Patients. Games Health J. 2016 Feb;5(1):27-33. doi: 10.1089/g4h.2015.0001. Epub 2015 Nov 18. PMID 26579590
- [Result] Cost-utility analysis of the telerehabilitation of heart patients : the Teledi@log project. / Kidholm, Kristian; Rasmussen, Maja Kjær; Andreasen, Jan Jesper; Hansen, John; Nielsen, Gitte; Dinesen, Birthe Irene. I: International Journal of Integrated Care, Vol. 15, Nr. ETC Conf. Suppl., 2015.
- [Result] Pedometer use as motivation for physical activity in cardiac tele-rehabilitation. / Thorup, Charlotte Brun; Grønkjær, Mette; Spindler, Helle; Andreasen, Jan Jesper; Hansen, John; Dinesen, Birthe Irene; Nielsen, Gitte; Sørensen, Erik Elgaard. I: International Journal of Integrated Care, Vol. 15, Nr. ETC Conf. Suppl., 2015.
- [Result] Telerehabilitation of cardiac patients : findings from an interdisciplinary telerehabilitation program. / Dinesen, Birthe Irene. I: Telemedicine and e-Health, Vol. 21, Nr. 5, 2015, s. A-59.
- [Result] Pedometer and physical activity for cardiac patients in a telerehabilitation program. / Thorup, Charlotte Brun; Andreasen, Jan Jesper; Dinesen, Birthe; Hansen, John; Grønkjær, Mette; Sørensen, Erik Elgaard. I: European Journal of Cardiovascular Nursing, Vol. 13, Nr. Suppl. 1, 2014, s. S17.
- [Result] Tværsektoriel kommunikationsplatform en gevinst i telerehabilitering af hjertepatienter på tværs af sektorer. / Skov, Christina; Sørensen, Stine Bæk; Dinesen, Birthe. 2014. Abstract from National Konference for Center for Innovativ Medicinsk Teknologi, CIMT, Middelfart, Danmark.
- [Result] Udvikling af Aktivthjerte.dk : en digital værktøjskasse til telerehabilitering af hjertepatienter i Teledi@log projektet via en brugerdreven innovations proces. / Dinesen, Birthe; Spindler, Helle. 2014. Abstract from National Konference for Center for Innovativ Medicinsk Teknologi, CIMT, Middelfart, Danmark.
- [Result] Heart patients' experiences and use of social media in their rehabilitation : a qualitative study. / Jørgensen, Camilla Bech; Hansen, John; Spindler, Helle; Andreasen, Jan Jesper; Nielsen, Gitte; Dinesen, Birthe. Scandinavian Conference on Health Informatics 2013, 20 August 2013, Copenhagen, Denmark. red. / Gustav Bellika; Ann Bygholm; Mette Dencker; Mariann Fossum; Gert Galster; Gunnar Hartvigsen; Ole Hejlesen; Daniel Karlsson; Sabine Koch; Carl-Erik Moe. Linköping University Electronic Press, 2013. s. 51-54 (Linköping Electronic Conference Proceedings; Nr. 91).
- [Result] Identification of heart patients' everyday need : Based on user-driven innovation. / Hæsum, Lisa Korsbakke Emtekær; Nielsen, G.; Hangaard, Stine Veje; Hejlesen, Ole; Dinesen, Birthe. Global Telemedicine and eHealth Updates : Knowledge Resources, 18-20 April 2012, Luxembourg. red. / Malina Jordanova; Frank Lievens. Vol. 5 International Society for Telemedicine & eHealth, 2012. s. 611-614 ( Global Telemedicine and eHealth Updates : Knowledge Resources, Vol. 5).
- [Result] Personal health record for chronic patient. / Dinesen, Birthe. The International eHealth, Telemedicine and Health ICT Forum for Education, Networking and Business, 18-20 April 2012, Luxembourg: Exhibition and Conference Guide. International Society for Telemedicine & eHealth, 2012. s. 123.
- [Derived] Dinesen B, Spindler H. The Use of Telerehabilitation Technologies for Cardiac Patients to Improve Rehabilitation Activities and Unify Organizations: Qualitative Study. JMIR Rehabil Assist Technol. 2018 Nov 19;5(2):e10758. doi: 10.2196/10758. PMID 30455168
- [Derived] Thorup C, Hansen J, Gronkjaer M, Andreasen JJ, Nielsen G, Sorensen EE, Dinesen BI. Cardiac Patients' Walking Activity Determined by a Step Counter in Cardiac Telerehabilitation: Data From the Intervention Arm of a Randomized Controlled Trial. J Med Internet Res. 2016 Apr 4;18(4):e69. doi: 10.2196/jmir.5191. PMID 27044310
- [Derived] Kidholm K, Rasmussen MK, Andreasen JJ, Hansen J, Nielsen G, Spindler H, Dinesen B. Cost-Utility Analysis of a Cardiac Telerehabilitation Program: The Teledialog Project. Telemed J E Health. 2016 Jul;22(7):553-63. doi: 10.1089/tmj.2015.0194. Epub 2015 Dec 29. PMID 26713491
- See also: Homepage for the study — http://teledialog.dk